CLINICAL TRIAL: NCT03463811
Title: Best Cutoff Value of Lactate Concentration in Vaginal Fluid to Predict Time of Spontaneous Onset of Labor in PPROM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mennatallah Mohamed Elnemr (Other)
Responsible Party: Sponsor-Investigator, Mennatallah Mohamed Elnemr, Best Cutoff value of lactate concentration in vaginal fluid to predict time of spontaneous onset of labor in PPROM, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: MElnemr
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Aim is to Investigate Association Between Lactate Concentration in Vaginal Fluid and Time of Spontaneous Onset of Labor in PPROM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lactate concentration in vaginal fluid — Lactate concentration in vaginal fluid

SUMMARY:
The present study is aimed to assess whether lactate determination in vaginal fluid is associated with and can predict onset of labor for women with suspected preterm prelabor rupture of membranes (PPROMs).

DETAILED DESCRIPTION:
Study design: Prospective observational cohort

ELIGIBILITY:
Inclusion Criteria:

* Age 25-35 years old
* BMI 25-30
* Singleton pregnancy in presentation with a history of suspected PPROM
* A live fetus with gestational age between 26+0 weeks and 34+0 weeks

Exclusion Criteria:

* Abruption placenta
* Medical disorders and hypertensive disorders of pregnancy
* Intrauterine fetal death
* Known or suspected fetal anomalies
* Signs of infection (Fever, increase total leucocytic count)
* Multiple pregnancy.
* Regular uterine contractions.
* History of cervical insufficiency

Ages: 25 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: This study will be conducted on 42 healthy pregnant with preterm PROM women they will be investigated for lactate concentration in vaginal fluid and observed for latency period till onset of spontaneous labor
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Time from examination to spontaneous onset of labor | 48 hours
  Time from examination to spontaneous onset of labor < or > 48 hours according to concentration of lactate in vaginal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khairy, prof, Study Director — Ainshams university
Locations (1):
- Ain shams, Cairo, Egypt